CLINICAL TRIAL: NCT05484232
Title: Outcomes of Early Laparoscopic Cholecystectomy in Cases of Acute Cholecystitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sherif Ali Ahmed, resident doctor at general surgery department at sohag university, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-07-10
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Acute Calculous Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Early laparoscopic cholecystectomy in patients with acute calcular cholecystitis

SUMMARY:
Laparoscopic cholecystectomy is the most common laparoscopic surgery performed in the world. The initial treatment of acute calculus cholecystitis includes GIT rest, intravenous fluid, correction of electrolyte imbalance from repeated vomiting, good analgesia, and intravenous antibiotics. Following this treatment, patients with uncomplicated disease are managed on outpatient basis and are called for elective laparoscopic cholecystectomy after a period of 6-8 weeks.

Elective laparoscopic cholecystectomy has become the gold standard for treatment of symptomatic gallstones. However, in the early days, acute cholecystitis was a contraindication of laparoscopic cholecystectomy, and patients with acute cholecystitis were managed conservatively and discharged for re-admission in order to have elective surgery performed for the definitive treatment.

Early laparoscopic cholecystectomy, within 72 hours of presentation,has been advocated because of shorter hospital stay, decreased financial costs and reduced readmission rates. Previously cited reasons against early laparoscopic cholecystectomy include the increased technical difficulties, increased risk of conversion to an open procedure (6-35 % in some studies) and increased risks of biliary complications such as bile leaks and common bile duct (CBD) injuries when operating on an inflamed gallbladder with edematous planes and distorted anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presented by Acute cholecystitis fit for lap cholecystectomy .

Exclusion Criteria:

* Patients unfit for laparoscopic surgery such as patients with significant medical illness (ASAgrade more 3), pancreatitis and common bile duct stones

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
duration of surgery , | Intraoperative
  compare between duration of surgery between traditional elective laparoscopic cholecystectomy and early laparoscopic cholecystectomy
percentage of complications | 6 months
  compare between percentage of complications of surgery between traditional elective laparoscopic cholecystectomy and early laparoscopic cholecystectomy
morbidity | 6 months
  compare morbidity between traditional elective laparoscopic cholecystectomy and early laparoscopic cholecystectomy
mortality | 6 months
  compare mortality between traditional elective laparoscopic cholecystectomy and early laparoscopic cholecystectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gul R, Dar RA, Sheikh RA, Salroo NA, Matoo AR, Wani SH. Comparison of early and delayed laparoscopic cholecystectomy for acute cholecystitis: experience from a single center. N Am J Med Sci. 2013 Jul;5(7):414-8. doi: 10.4103/1947-2714.115783. PMID 24020050
- [Background] Ozkardes AB, Tokac M, Dumlu EG, Bozkurt B, Ciftci AB, Yetisir F, Kilic M. Early versus delayed laparoscopic cholecystectomy for acute cholecystitis: a prospective, randomized study. Int Surg. 2014 Jan-Feb;99(1):56-61. doi: 10.9738/INTSURG-D-13-00068.1. PMID 24444271
- [Background] Cao AM, Eslick GD, Cox MR. Early Cholecystectomy Is Superior to Delayed Cholecystectomy for Acute Cholecystitis: a Meta-analysis. J Gastrointest Surg. 2015 May;19(5):848-57. doi: 10.1007/s11605-015-2747-x. Epub 2015 Mar 7. PMID 25749854
- [Background] Minutolo V, Licciardello A, Arena M, Nicosia A, Di Stefano B, Cali G, Arena G. Laparoscopic cholecystectomy in the treatment of acute cholecystitis: comparison of outcomes and costs between early and delayed cholecystectomy. Eur Rev Med Pharmacol Sci. 2014 Dec;18(2 Suppl):40-6. PMID 25535191